CLINICAL TRIAL: NCT03882385
Title: Screening For Critical Congenital Anomalies In NICU And Their Out Come in Assiut Universty
Brief Title: Screening For Critical Congenital Anomalies In NICU And Their Out Come
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Tharwat Helmy, principal investigator, Assiut University
Other Study IDs: SCCAS
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Congenital Anomaly
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The congenital malformation (CMF) include disturbance in normal process of organogenesis occurring before birth .

* The (CMF) are structural ,functional, or (biochemical Molecular) defect presenting at birth.
* The structural defect resulting from prenatal insult during period of embryogeneses.
* The neonate with congenital malformation have differences in physiology, anatomy, in response to stress.
* The (CMF) are important causes of infant disability , illness, deaths.
* (CMF) classified into mild, moderate, severe and lethal

DETAILED DESCRIPTION:
The (CMF) may be structural abnormalities with significant effect on function (e.g) cleft palate .

Or minimal effect on clinical function but may have cosmotic impact (e.g) pre-auricular pit .

In developed countries, outcome of neonatal congenital anomalies is favourable because of availability of antenatal diagnosis, improved surgical skills and technologies, sophisticated neonatal intensive care unit, availability of total parenteral nutrition and adequate staff.

In developing countries, however, neonatal surgery is still fraught with a lot of problems including late presentation and lack of medical facilities and human resources, thereby, making newborn surgery to be associated with unacceptably high morbidity and mortality.

Due to the burden of other neonatal and childhood diseases in developing countries, neonatal surgery is often considered low priority in healthcare budget planning and allocation.

* Effective live , saving medical treatment is available for survival birth defects with functional disorders .
* Neonatal with birth defect may be further referred to appropriate level of medical , surgical facilities .

Risk factors:

* Unknown cause
* Preconception causes are genetic and partially genetic, originating mostly before conception. Birth defects are due to abnormalities of the genetic material-chromosomes and genes including chromosomal abnormalities, single gene defects and multifactorial disorders (which are caused by the interaction of genes and the environment).
* Post-conception causes develop after conception, but before birth. Birth defect is caused by an intra-uterine environmental factor. This includes teratogens that interfere with normal growth and development of the embryo or foetus, mechanical forces that deform the foetus, and vascular accidents that disrupt the normal growth of organs.
* Socioeconomic and demographic factors:

Congenital anomalies are more frequently seen among low income families and countries.

* Maternal age: advanced maternal age increases the risk of chromosomal abnormalities, such as Down syndrome.
* Infections:

Some Maternal infections during pregnancy can increase the risk of birth defects such as:

Rubella infection (German measles-a viral infection) to pregnant mother can result in to miscarriage, deafness, intellectual disability, heart defects and blindness in newborn.

Toxoplasmosis (disease caused by parasite found in soil) infection during pregnancy can cause birth defects such as hearing loss, vision problems and intellectual disability.

Sexually transmitted infections (STIs): such as syphilis, cytomegalovirus can cause serious birth defects.

Zika virus infection: during pregnancy can cause certain birth defects (microcephaly and other abnormalities).

• Environmental factors: Maternal exposure to certain medications, psychoactive drugs, tobacco, radiation and pesticides during pregnancy may increase the risk of congenital anomalies in foetus or neonate.

Working or living near, or in, waste sites, smelters or mines may also be a risk factor.

Certain drugs when taken during pregnancy may cause birth defects; these drugs are called teratogenic drugs (Category 'X' drugs). Categories 'X' drugs are contraindicated during pregnancy. (Drugs are categorized into 5 categories according to the development of adverse effects on the foetus, category A, B, C, D and X.)

ELIGIBILITY:
Inclusion Criteria:

* • Cases need resustation and stabilization.

  * Congenital anomalies that need admission in NICU eg: impeforated anus , meningiocele, heart disease, tacho osphageal fistula, urinary problems, diaphragmatic hernia, intestinal obstruction, duedodnal obstruction, neural tube defect .

Exclusion Criteria:

* All vitally stable cases that don't need NICU admission and all cases not need immediate intervention of congenital anomalies

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: study on neonates born with critical congenital anomalies that need intervention in NICU need resuscitation or refere to other specialist
Sampling Method: Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2019-03-19 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-11-29 (Estimated)

PRIMARY OUTCOMES:
detect number of total babies and percentages of congenital anomalies | 24 hours

REFERENCES:
- [Background] Bassil KL, Collier S, Mirea L, Yang J, Seshia MM, Shah PS, Lee SK; Canadian Neonatal Network. Association between congenital anomalies and area-level deprivation among infants in neonatal intensive care units. Am J Perinatol. 2013 Mar;30(3):225-32. doi: 10.1055/s-0032-1323584. Epub 2012 Aug 9. PMID 22879358